CLINICAL TRIAL: NCT01694862
Title: Integra Initiative to Assess the Benefits and Costs of Integrating Sexual and Reproductive Health and HIV Services in Kenya and Swaziland
Brief Title: Benefits and Costs of Integrating Sexual-Reproductive Health and HIV Services in Kenya and Swaziland
Acronym: Integra
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Population Council (Other); International Planned Parenthood Federation (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Susannah Mayhew, Reader (Professor), London School of Hygiene and Tropical Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Integra Initiative
Record Dates: First submitted 2012-09-21; First posted 2012-09-27 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Pregnancy; HIV
Keywords: quasi experimental; evaluation; intervention; service integration; cost analysis; HIV; FP; PNC; Sub-Saharan Africa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrated FP /PNC service delivery (Experimental): Clinic or district identified as 'intervention' in which FP and PNC services are (theoretically) being provided together with HIV services (counselling, testing, treatment etc.) and in which the procedural intervention has been applied.
  Interventions: Procedure: Integrated FP/PNC service delivery
- Non-integrated FP/PNC service delivery (No Intervention): Clinic or district where FP and PNC services are not (theoretically) being provided together with HIV services, and in which no procedural intervention has been applied.

INTERVENTIONS:
Procedure: Integrated FP/PNC service delivery — The intervention uses a procedural tool building on existing MoH procedures. It has nine components: strengthening protocols, guidelines and training materials for integrated HIV-SRH care; training, mentorship; developing a mentoring and supervisory package; improving provider capacity; ensuring availability of minimum levels of equipment and supplies for integrated services; support supervision; organizational change (including reviewing use of available rooms) and role clarification; improving availability of IEC/BCC materials on FP and HIV; strengthening the referral system between FP and ART and the data collection and recording systems.
  Other Names: BCS+
  Arms: Integrated FP /PNC service delivery

SUMMARY:
The overarching aim of the Integra Initiative is to strengthen the evidence base on the impact of integrating family planning (FP), postnatal care (PNC) and HIV services in sub-Saharan Africa. Specifically, in the study the investigators aim to test the following hypotheses:

the provision of integrated services, compared to separate services, will:

1. lead to increased uptake of a range of SRH services .
2. attract a greater number and diversity of clients.
3. lead to increased quality of a range of SRH services
4. lead to healthier sexual and reproductive behavior.
5. lead to reduced stigma at health facilities.
6. lead to the more efficient use of resources, with a lower unit cost of provision of key services.

For the purposes of this study integration is defined as offering clients both HIV and postnatal care (PNC) or HIV and family planning (FP) services in the same visit.

To better understand how services can be integrated in different countries this study focuses on two key models of integration in Kenya and Swaziland.

* The first model focuses on integration of FP and HIV services (integrated FP model) and entails performing HIV testing, STI screening and management, cervical cancer screening, condom promotion within FP consultations, as well as active referral to antiretroviral (ART) units for HIV-positive clients. The FP model will be evaluated in Kenya only.
* The second model focuses on integration of PNC and HIV services (integrated PNC model) and will be implemented in both Kenya and Swaziland. The model focuses on the provision of PNC services to mother and baby, FP services, repeat HIV testing for mother, HIV testing for infant and referral to HIV services for HIV positive mothers and infants, as well as referrals for clients requiring other additional services.

DETAILED DESCRIPTION:
There are many well-established reasons that support the rationale for integrating or linking sexual and reproductive health (SRH) and HIV services in developing countries with generalized HIV epidemics - primarily in sub-Saharan Africa. Yet the evidence base for the impact of integrated service delivery on health outcomes and costs remains weak. Partly this is a result of methodological difficulties.

There is an emerging body of literature addressing the challenges of using randomized controlled trials to assess the impact of public health interventions. Particularly in cases such as the Integra Initiative, where the causal chain (between intervention and outcome) is long, and where there are is a broad range of outcomes that need to be explored, and where there is already some a degree of integration occurring in some clinic settings, attempting to conduct a randomized controlled trial is not appropriate. Consistent with evaluation designs described by Habicht and colleagues, the Integra design includes evaluation of performance and impact to try to make two types of causal inference: adequacy and plausibility.

Evaluation of adequacy will assess whether the expected changes in provision, service utilisation and cost-effectiveness have occurred in intervention facilities. Evaluation of impact will assess the plausibility that changes in service, health and behavioral outcomes are due to the Integra Initiative. The case for such plausibility will be built from the following strands of evidence:

* Comparing findings in 'intervention' facilities with those in facilities chosen as 'comparison' sites prior to the evaluation
* Exploring a dose-response relationship between the measured extent of integration and the study outcomes
* Measuring changes in performance over time, to demonstrate a logical sequence between the intervention (integration) and outcomes.
* Measuring change in each step of the logic model - a prerequisite for any attribution to the intervention
* Triangulating findings from a mix of research methods to capture a range of perspectives and insights from different disciplines.

The study will employ a controlled pre- and post-test quasi-experimental, or non-randomised, design and utilises multiple research methods (cohort study, community survey, clinic assessments, costing tools and qualitative interviews). Since the research is being conducted in real-life health delivery settings where programmatic contamination is possible due to ongoing health programme interventions over the study period, the control group will be referred to as a 'comparison group', for which outcomes will be compared over time up to two years after implementation.

ELIGIBILITY:
Inclusion Criteria for FP-HIV study:

* women aged 15 years and over,
* be revisit FP clients,
* be living in the catchment area of the health facility, and
* willing to give their informed consent to be interviewed.

Inclusion Criteria for PNC-HIV study:

* women aged 15 years and over,
* be postnatal clients attending a postnatal check for themselves and/or their infant (0-10 weeks),
* living in the catchment area of the health facility, and
* willing to give their informed consent to be interviewed.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4763 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Unintended pregnancies | 24 months
  Unintended pregnancy measures:
  * percent women who become pregnant (cohort study)
  * percent HIV+/HIV- women reporting planned pregnancy (cohort and client exit interviews)
  * percent clients women with correct knowledge of fertile period (cohort, client exit interviews) Proportion of population who report unintended pregnancy in last 12 months (community survey)

SECONDARY OUTCOMES:
HIV risk behaviour | 24 months
  HIV risk measures:
  * Condom use at last sex (cohort, client exit interviews, community survey)
  * Number of partners in past 12 months (cohort, client exit interviews, community survey)
  * Received STI/HIV counseling (cohort, client exit interviews, community survey) Consistent condom use reported (cohort, client exit interviews, community survey)
  * Use of condoms with another FP method (dual protection )(cohort, client exit interviews, community survey)

OTHER OUTCOMES:
Unit costs | 24 months
  Economics measures in 42 study clinics:
  * Cost per eligible client receiving ART,
  * Cost per person-month of receiving ART
  * Cost per client counseled, tested and receiving results
  * Cost per client receiving each service component

CONTACTS AND LOCATIONS:
Overall Officials: Susannah H Mayhew, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (2):
- Multiple MoH locations in Swaziland, Manzini, Eswatini
- Multiple MoH facilities in Kenya, Thika, Nyeri and Others, Kenya

REFERENCES:
- [Derived] Birdthistle IJ, Fenty J, Collumbien M, Warren C, Kimani J, Ndwiga C, Mayhew S; Integra Initiative. Integration of HIV and reproductive health services in public sector facilities: analysis of client flow data over time in Kenya. BMJ Glob Health. 2018 Sep 14;3(5):e000867. doi: 10.1136/bmjgh-2018-000867. eCollection 2018. PMID 30245866
- [Derived] Wekesa E, Askew I, Abuya T. Ambivalence in pregnancy intentions: The effect of quality of care and context among a cohort of women attending family planning clinics in Kenya. PLoS One. 2018 Jan 9;13(1):e0190473. doi: 10.1371/journal.pone.0190473. eCollection 2018. PMID 29315327
- [Derived] Mayhew SH, Colombini M, Kimani JK, Tomlin K, Warren CE; Integra Initiative; Mutemwa R. Fertility intentions and contraceptive practices among clinic-users living with HIV in Kenya: a mixed methods study. BMC Public Health. 2017 Jul 5;17(1):626. doi: 10.1186/s12889-017-4514-2. PMID 28679389
- [Derived] Kimani J, Warren CE, Abuya T, Ndwiga C, Mayhew S, Vassall A, Mutemwa R, Askew I. Use of HIV counseling and testing and family planning services among postpartum women in Kenya: a multicentre, non-randomised trial. BMC Womens Health. 2015 Nov 13;15:104. doi: 10.1186/s12905-015-0262-6. PMID 26563220
- [Derived] Obure CD, Guinness L, Sweeney S, Initiative I, Vassall A. Does integration of HIV and SRH services achieve economies of scale and scope in practice? A cost function analysis of the Integra Initiative. Sex Transm Infect. 2016 Mar;92(2):130-4. doi: 10.1136/sextrans-2015-052039. Epub 2015 Oct 5. PMID 26438349
- [Derived] Kimani J, Warren C, Abuya T, Mutemwa R; Integra Initiative; Mayhew S, Askew I. Family planning use and fertility desires among women living with HIV in Kenya. BMC Public Health. 2015 Sep 17;15:909. doi: 10.1186/s12889-015-2218-z. PMID 26381120
- [Derived] Mulrenan C, Colombini M, Howard N, Kikuvi J, Mayhew SH; Integra Initiative. Exploring risk of experiencing intimate partner violence after HIV infection: a qualitative study among women with HIV attending postnatal services in Swaziland. BMJ Open. 2015 May 14;5(5):e006907. doi: 10.1136/bmjopen-2014-006907. PMID 25976760
- [Derived] Birdthistle IJ, Mayhew SH, Kikuvi J, Zhou W, Church K, Warren CE, Nkambule R, Fenty J; Integra Initiative. Integration of HIV and maternal healthcare in a high HIV-prevalence setting: analysis of client flow data over time in Swaziland. BMJ Open. 2014 Mar 7;4(3):e003715. doi: 10.1136/bmjopen-2013-003715. PMID 24607560
- [Derived] Warren CE, Mayhew SH, Vassall A, Kimani JK, Church K, Obure CD, du-Preez NF, Abuya T, Mutemwa R, Colombini M, Birdthistle I, Askew I, Watts C. Study protocol for the Integra Initiative to assess the benefits and costs of integrating sexual and reproductive health and HIV services in Kenya and Swaziland. BMC Public Health. 2012 Nov 13;12:973. doi: 10.1186/1471-2458-12-973. PMID 23148456
- See also: Project website — http://www.integrainitiative.org/